CLINICAL TRIAL: NCT00034203
Title: Safety and Efficacy of a Monoclonal Antibody for Treatment of Rheumatoid Arthritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: HURA501
Record Dates: First submitted 2002-04-23; First posted 2002-04-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — efalizumab

INTERVENTIONS:
Drug: efalizumab

SUMMARY:
The purpose of this study is to determine whether a humanized monoclonal antibody (efalizumab) is safe and effective in the treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of moderate to severe rheumatoid arthritis.
* On stable dose of methotrexate.
* 18 to 80 years of age.
* Less than 275 lbs.

Exclusion criteria:

* Joint replacement surgery within 60 days of the start of drug dosing.
* Intra-articular cortisone injections within 28 days of the start of drug dosing.
* Pregnancy.
* History of severe allergic or anaphylactic reactions.
* Active bacterial, viral, fungal, mycobacterium tuberculosis.
* Positive PPD test.
* History of any opportunistic infection.
* Serious persisting local or systemic infection.
* History of malignancy within the past five years.
* Received any vaccine within 28 days of the start of study drug dosing.
* Joint replacement therapy planned within nine months of the start of study drug dosing.
* Chronic disorders apart from RA affecting the joints.
* Significant systemic involvement secondary to RA.
* COPD, asthma, or other pulmonary disease.
* Received any DMARD other than methotrexate in the 28 days prior to the start of study drug dosing.
* Approved biologic RA therapy during the 28 days or 7 half-lives of the drug prior to the start of drug dosing.
* Investigational drug and/or treatment during the 28 days or seven half-lives of the investigational drug prior to the start of study drug dosing.
* Liver disease or abnormal hepatic function.
* Serum creatinine level > 1.5 mg/dL.
* Platelet count < 125,000 cells/mm3.
* WBC count < 3,500 cells/mm3.
* Seropositive for hepatitis B surface antigen.
* Seropositive for hepatitis C antibody.
* Known seropositivity for HIV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (52):
- United States (52):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Arizona Arthritis Research, PLC, Paradise Valley, Arizona
  - Advanced Clinical Therapeutics, LLC, Tucson, Arizona
  - NEA Clinic, Jonesboro, Arkansas
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - University of California at San Diego, La Jolla, California
  - UCLA, Los Angeles, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - Desert Medical Advances, Rancho Mirage, California
  - The San Diego Arthritis and Osteoporosis Medical Clinic, San Diego, California
  - Pacific Arthritis Center, Santa Maria, California
  - Northeast Clinical Research, LLC, Hamden, Connecticut
  - Clinical Research Consultants, Inc., Trumbull, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - The Center for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Anchor Research Center, Naples, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - nTouch Research Corporation, St. Petersburg, Florida
  - Tampa Medical Group, Tampa, Florida
  - nTouch Research Corporation, Vero Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - nTouch Research Corporation, Decatur, Georgia
  - nTouch Research Corporation, Marietta, Georgia
  - Tri-State Arthritis and Rheumatology Center, LLC, Evansville, Indiana
  - Central Iowa Hospital Corporation, Des Moines, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Phase III Clinical Research, Fall River, Massachusetts
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Washington University Center for Clinical Studies, St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Bassett Healthcare Clinical Pharmacology Research Center, Cooperstown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Hospital for Joint Disease, ACRC, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Prem C. Chatpar, M.D., Plainview, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - McBride Clinic, Inc., Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - nTouch Research Corporation, Pittsburgh, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Volunteer Research Group, LLC, Knoxville, Tennessee
  - Summit Research Solutions, Inc., Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Austin Rheumatology Research, Austin, Texas
  - Physicians' Research Options, LLC, Ogden, Utah
  - South Puget Sound Clinical Research, Olympia, Washington
  - University of Wisconsin, Madison, Madison, Wisconsin